## Statistical Analysis Plan

Study Title: "Facebook and Friends" Developing an Effective Online Social Network for Weight Loss

NCT02656680

We summarized engagement, retention, and acceptability using descriptive statistics. For variables that were normally distributed, we described distributions using mean and standard deviation (M[SD]), and for variables that were not normally distributed, we described distributions using median and inter-quartile range (IQR). We compared retention and acceptability by treatment condition using chi-squared tests, or Fisher's exact tests as appropriate. We compared treatment conditions on engagement using a Wilcoxon rank-sum test. All randomized participants were included in the weight analyses except for 1 participant who became pregnant during the study. For participants who did not provide weight at follow-up, we also used their baseline weight.